CLINICAL TRIAL: NCT03706937
Title: The Treatment of Addictions in the Course of Care in Oncology: an Inventory of Fixtures Among Paramedical Professionals
Acronym: PREFACE
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1001
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Paramedical Professional
Keywords: Addiction; Tobacco; Oncology; Care pathways; Motivational attitude; Motivational interviewing; Nursing
MeSH Terms: conditions — Behavior, Addictive; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paramedical professionals: Paramedical professionals of the Lucien Neuwirth Cancer Institute
  Interventions: Other: Semi directive interview

INTERVENTIONS:
Other: Semi directive interview — Semi directive interview will be performed to try to define the management of addictions in the oncology care course. Thus, an approach in terms of social representations among paramedical professional actors involved in the care of patients treated for cancer and with an unresolved addictive disorder sounds the best way for this research.

SUMMARY:
Nowadays, guidance is given on the implementation of innovative approaches to promote autonomy and user participation through strategies designed to strengthen the patient's empowerment. [SNS 2018-2022, Ministère des Solidarités et de la Santé] The 2014-2019 Cancer Plan calls for the systematic support of smokers during smoking cessation. This means that health workers need to be trained to help with smoking cessation, as well as the motivational attitude that reinforces the patient's smoker's self-esteem as well as his desire to off-load this addiction. [Perriot, Underner, Peiffer, Dautzenberg, 2018] It is recommended that these interventions be included from the beginning of the management, once the diagnosis of Cancer is made. It seems legitimate then to wonder about the place of choice the Motivational Interview (EM) could have in the course of cancer care, for the management of addictions during the treatment of cancer. We therefore wish to carry out descriptive qualitative research in the Lucien Neuwirth Oncology Institute in order to try to define the management of addictions in the oncology care course. Thus, an approach in terms of social representations among paramedical professional actors involved in the care of patients treated for cancer and with an unresolved addictive disorder sounds the best way for this research.

DETAILED DESCRIPTION:
Nowadays, guidance is given on the implementation of innovative approaches to promote autonomy and user participation through strategies designed to strengthen the patient's empowerment. [SNS 2018-2022, Ministère des Solidarités et de la Santé] The 2014-2019 Cancer Plan calls for the systematic support of smokers during smoking cessation. This means that health workers need to be trained to help with smoking cessation, as well as the motivational attitude that reinforces the patient's smoker's self-esteem as well as his desire to off-load this addiction. [Perriot, Underner, Peiffer, Dautzenberg, 2018] It is recommended that these interventions be included from the beginning of the management, once the diagnosis of Cancer is made. It seems legitimate then to wonder about the place of choice the Motivational Interview (EM) could have in the course of cancer care, for the management of addictions during the treatment of cancer. We therefore wish to carry out descriptive qualitative research in the Lucien Neuwirth Oncology Institute in order to try to define the management of addictions in the oncology care course. Thus, an approach in terms of social representations among paramedical professional actors involved in the care of patients treated for cancer and with an unresolved addictive disorder sounds the best way for this research.

ELIGIBILITY:
Inclusion Criteria:

- voluntary participation of health professionals in the Lucien Neuwirth Cancer Institute

Exclusion Criteria:

- refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Paramedical professional actors involved in the care of patients treated for cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of addiction managements | 3 months
  We therefore wish to carry out descriptive qualitative research in the Lucien Neuwirth Oncology Institute in order to try to define the management of addictions in the oncology care course. In a first time, number of addiction managements will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Verot, Study Director — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verot E, Regnier Denois V, Macron C, Chauvin F. Managing unresolved issues of addiction during cancer treatment: A qualitative study about cancer care providers' representations. PLoS One. 2020 Nov 24;15(11):e0242693. doi: 10.1371/journal.pone.0242693. eCollection 2020. PMID 33232348